CLINICAL TRIAL: NCT02893098
Title: A Study to Evaluate the Safety and Efficacy of Humia Inj. in Patients With Symptomatic Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Huons Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HU-025 P3
Record Dates: First submitted 2016-08-17; First posted 2016-09-08 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Osteoarthritis of Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Humia inj. (Experimental): Participants with symptomatic Primary Osteoarthritis of Knee received a single injection of 3ml Humia inj.
  Interventions: Drug: Humia inj.
- High Hyal Plus inj. (Active Comparator): Participants (Control Group) with symptomatic Primary Osteoarthritis of Knee received single injection of 2ml High Hyal Plus inj. given weekly for 3 weeks
  Interventions: Drug: High hyal Plus inj.

INTERVENTIONS:
Drug: Humia inj. — Single injection of 3mL Humia inj.
  Dummy: Single injection 2ml Normal Saline inj. given weekly for 2 weeks
  Arms: Humia inj.
Drug: High hyal Plus inj. — Single Injection of 2mL High hyal Plus inj. given weekly for 3 weeks
  Arms: High Hyal Plus inj.

SUMMARY:
A Multi-Centre, Parallel, Double-Blind, Active comparator, Randomised phase III Clinical Trial

ELIGIBILITY:
Inclusion Criteria:

* Primary knee osteoarthritis confirmed clinically and radiologically according to American College of Rheumatology criteria have joint pain
* Kellgren-Lawrence Grade Ⅰ to Ⅲ confirmed radiologically within 6 months
* Knee pain under weight-bearing pain(100mm-VAS) greater than 40mm
* Able to walk without assistive devices
* Patients willing and able to provide signed informed consent after the nature of the study has been explained

Exclusion criteria:

* Body Mass Index (BMI) > 32
* History of rheumatoid arthritis or other inflammatory arthritis in knee articular cavity
* Systemic Intravenous Steroid injection within 1 month, intra-articular corticosteroid injection within 3 months or hyaluronate injection within 6 months
* Has clinically severe tense effusion of the target knee diagnosed Positive according to Patella tap test
* Undergo Knee Replacement Surgery of the target knee

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-10 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline of Weight-bearing pain (100mm-VAS) | Week 14

SECONDARY OUTCOMES:
Change from baseline of Weight-bearing pain (100mm-VAS) | Weeks 3, 8, 14, and 26
Change from Visit 8 of Weight-bearing pain (100mm-VAS) | Week 38
Physical Examination : Swelling | Weeks 0, 3, 8, 14, 26, and 38
Physical Examination : Tenderness on pressure | Weeks 0,3,8,14,26,and 38
Physical Examination : Range of motion | Weeks 0, 3, 8, 14, 26, and 38
Consumption of rescue medication | Weeks 0, 1, 2, 3, 8, 14, 26, and 38
Proportion (%) of patients taking rescue medication | Weeks 0, 1, 2, 3, 8, 14, 26, and 38
Responder Rate | Week 14

CONTACTS AND LOCATIONS:
Locations (1):
- Huons, Ansan-si, Gyeonggi-do, South Korea